CLINICAL TRIAL: NCT02988102
Title: Role of Concentration of Biomarkers S100B and NSE in Serum in Mild and Moderate Head Trauma Injury in Acute Phase in Relation to Head CT and Post Concusion Syndrome.
Brief Title: Role of Concentration of Biomarkers S100B and NSE in Serum in Mild and Moderate Head Trauma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Clinical Centre of Kosova (Other)
Responsible Party: Principal Investigator, Dr. Fatos Kelmendi, Dr. Fatos Kelmendi Neurosurgeon, University Clinical Centre of Kosova
Other Study IDs: FKelmendi
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Biomarkers
Keywords: S100B, NSE; moderate brain trauma; mild brain trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biomarkers S100B and NSE in blood sample ( Venous blood)
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Following S100B and NSE in head trauma — Following S100B and NSE in head trauma in correlation with Head CT and post concussion syndrome and Lisat11
  Other Names: S100B NSE

SUMMARY:
In pediatric age groups communication difficulties very sometimes may present further obstacles in obtaining a detailed injury history and early identification of TBI symptoms.

Most emergency management protocols are focused exclusively on the identification of the relatively small number of patients who may require operative intervention, as early surgery is believed to improve outcome.

DETAILED DESCRIPTION:
However early rehabilitation can also be effective for the much larger number of patients who do not require surgery[1] In addition, Hall and others recently reported that low doses of ionizing radiation to the brain in infancy may influence cognitive abilities in adulthood. [2] Accordingly, increased serum concentrations of, for example S100B ( a calcium-binding protein present in high concentrations in glial cells) and neurone-specific enolase ( NSE: a cytoplasmatic enzyme occuring predominantly in neurones ) have been demonstrated to reflect the presence and severity of brain tissue damage in acute head injuries. [3] In both pediatric age and adults.

ELIGIBILITY:
Inclusion Criteria:

* Only head trauma without any other body injury

Exclusion Criteria:

* Blood thinner, hydrocephalus , previous brain infarcts, encephalopathy, birth trauma.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 2 groups pediatric and adult.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2016-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Role of concentration of biomarkers S100B and NSE in serum in mild and moderate head trauma injury in acute phase in relation to head CT and post concusion syndrome. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fatos Kelmendi, Tirana, Kosovo Prishtina, Albania

IPD SHARING:
Plan to Share IPD: No